CLINICAL TRIAL: NCT05477537
Title: Adapted Physical Activity in the Treatment of Anorexia:
Acronym: EfAPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Santé des Étudiants de France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A00416-37
Record Dates: First submitted 2022-07-22; First posted 2022-07-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa
Keywords: Adapted physical activity
MeSH Terms: conditions — Anorexia Nervosa | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This protocol is to carry out an open, multi-centric, randomized controlled trial assessing a population of adolescents suffering from Anorexia Nervosa according to the DSM-5 criteria.
  Randomisation will be centralised and stratified according to the status of treatment at inclusion (ambulatory care or day hospitalisation - the latter possibly entailing a selection bias for reason of severity), and the centre. A randomisation list will be generated on computer with blocks of variable size by a statistician independent from the group recruiting or taking care of patients at INSERM CESP, it will be include in the e-CRF procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Add-on group (Experimental): Subjects with Anorexia Nervosa (AN) involved in a day hospital or an inpatient program following HAS guidelines for anorexia nervosa treatment (treatment as usual) who will receive in addition an adapted physical activity program (one lesson per week, during 8 weeks)
  Interventions: Other: Adapted physical activity program
- Treatment as usual group (Active Comparator): Subjects with Anorexia Nervosa involved in a day hospital or an inpatient program following HAS guidelines for AN treatment (treatment as usual).
  Interventions: Other: Treatment as usual group

INTERVENTIONS:
Other: Adapted physical activity program — subjects with Anorexia Nervosa (AN) involved in a day hospital or an inpatient program following HAS guidelines for anorexia nervosa treatment (treatment as usual) who will receive in addition an adapted physical activity program (one lesson per week, during 8 weeks) Adapted Physical Activity program, including psychoeducation on both problematic physical activity and consequences in terms of physical activity good practice leads to a better outcome among persons suffering from anorexia nervosa.
  Other Names: APA
  Arms: Add-on group
Other: Treatment as usual group — Subjects with Anorexia Nervosa involved in a day hospital or an inpatient program following HAS guidelines for AN treatment (treatment as usual)
  Arms: Treatment as usual group

SUMMARY:
People with anorexia nervosa are known to engage in significant physical activity or sports. This practice is problematic because of the state of malnutrition, its interference with re-nutrition and the somatic and nutritional complications that the effect of physical activity can cause in these people. This significant physical activity is also called hyperactivity in the literature, it is in fact a problematic use of physical activity, it is a symptom commonly observed in people suffering from anorexia nervosa (in 31 to 80% cases).

In this context, Ms. Kern lecturer in Sciences and Techniques of Physical and Sports Activities (STAPS) at the University of Paris Nanterre has developed in collaboration with the clinical team (Pre Godart) an adapted physical activity program (APA) , for patients suffering from anorexia nervosa. The APA program includes 8 sessions of 1h30 including an important part of psychoeducation. The effectiveness of this program will be evaluated in terms of both restoration of body mass index and improvement in overall health.

The project's hypothesis is that adding a standardized 8-week Adapted Physical Activity program to the usual care, including psychoeducation on both problematic physical activity and the consequences in terms of good practice of physical activity leads to a better outcome of overall care in people with anorexia nervosa.

DETAILED DESCRIPTION:
The project's hypothesis is adding an 8 weeks standardized Adapted Physical Activity program, including psychoeducation on both problematic physical activity and consequences in terms of physical activity good practice leads to a better outcome among persons suffering from anorexia nervosa.

Expected consequences of the study: demonstration that including adapted physical activity program in the global treatment program of anorexia nervosa is crucial in order to improve the therapeutic efficacy of the treatment acceptability, as drop out is usually important. In case of positive results, it will allow suppress interdiction in doing sport, source of conflict - and a way to enhance compliance to treatment which is difficult in anorexia nervosa to enable greater, earlier efficacy, which is predictive of more rapid recovery and avoid of chronicity.

Main Objective To evaluate in terms of Body Mass Index evolution at the end of the program, the efficacy of a 8 weeks standardized adapted physical activity program, designed for persons suffering from anorexia nervosa, including psychoeducation on both problematic physical activity and consequences and in terms of physical activity good practices.

Secondary Objectives To evaluate, at the end and 6 months later, the efficacy of a 8 week standardized Adapted Physical Activity program (including psychoeducation in terms of physical activity good practices designed for persons suffering from anorexia nervosa on both problematic physical activity and consequences), in terms of variation of body composition evaluated by bioelectric impedance (Fat mass and fat free mass), physical activity (duration, intensity, addiction, compulsion), fitness perceived (general fitness, cardio respiratory, strength, agility, flexibility ), self-esteem , perception of the body shape, quality of life both in terms of general and specific and eating disorders symptoms, level of anxiety symptoms, level of depressive symptoms, level of eating disorders symptoms, rate of drop-out from the global treatment program. To evaluate also the variation of BMI between base line and 6 months, and between 8 weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia nervosa patients (DSM 5 criteria),
* over or equal to 12 years old,
* Treated in the specialised eating disorder centres involved in the study either in the day hospital program or in the inpatient program,
* Understanding, reading and writing French,
* Benefiting from social cover
* Have read the information notice and have consented to participate in the study by signing a written consent

Exclusion Criteria:

* Somatic instability needing intensive medical care or monitoring (intensity is adapted in each session to each patient) or psychiatric emergency (suicidal risk and/or acute psychiatric symptomatology),
* Somatic complication forbidding any physical activity,
* Absence social cover,
* Patients in an emergency situation, incapable of giving their consent or adults under guardianship or curatorship,
* Pregnant or breastfeeding women (declarative: question asked to the patient during inclusion),
* Refusal to participate.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index change | Inclusion (start of research) and 9 week later (=T3)
  Difference between the two groups (treatment as usual versus the add on group:ie: treatment as usual plus adapted physical activity) concerning the of change of body Mass Index (Weight/(height)² between baseline and the end of the adapted physical activity program (ie: at 8 weeks after baseline). Weight will be measured with the subject wearing only underwear on the same calibrated scales. Stature will be measured using a stadiometer.

SECONDARY OUTCOMES:
Physical self Change | First program session (T1= one week after inclusion) / 8 week later T1 (end of program = T2) / 6 month after T2 (=T4)
  Physical Self-inventory
Physical activity currently change | First program session (T1= one week after inclusion) / 8 week later T1 (end of program=T2) /6 month after T2 (=T4)
  Duration, intensity : Global Physical Activity Questionnaire (GPAQ)-
Physical activity currently change | First program session (T1= one week after inclusion) /8 week later T1 (end of program=T2) /6 month after T2 (=T4)
  Motivation for physical activity : Behavior Regulation Exercise Questionnaire (BREQ 3)
Physical activity currently change | First program session (T1= one week after inclusion) / 8 week later T1 (end of program=T2) / 6 month after T2 (=T4)
  Dependence : EXERCISE DEPENDENCE SCALE-REVISED (EDS-R)
Perception of the body shape change | First program session (T1= one week after inclusion) / 8 week later T1 (end of program=T2) / 6 month after T2 (=T4)
  Self questionnaire : Body Shape Questionnaire
Body image Matrix Of Thinness and Muscularity change | First program session (T1= one week after inclusion) / 8 week later T1 (end of program=T2) / 6 month after T2 (=T4)
  Self questionnaire : Body image Matrix Of Thinness and Muscularity
Quality of life change | First program session (T1= one week after inclusion) / 8 week later T1 (end of program=T2) / 6 month after T2 (=T4)
  Self questionnaire : World Health Organization Quality of Life (Whoqol)
Anxiety and depression symptoms and stress change | First program session (T1= one week after inclusion) / 8 week later T1 (end of program=T2)
  Psychometric properties of the Depression Anxiety Stress Scales (EDAS)
Eating disorders symptoms change | Inclusion (start of research) and 8 month after inclusion
  Eating Disorder Examination Questionnaire (EDE-Q)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Godart, PU-PH, Study Director — Fondation Santé des Étudiants de France
Locations (7):
- France (7):
  - CHU Lille, Lille
  - Clinique Saint Vincent de Paul, Lyon
  - CHU Montpellier, Montpellier
  - CHU Nantes - service d'addictologie et Psychiatrie de Liaison, Nantes
  - GHU Saine Anne, Paris
  - UDJ Michel Ange, Paris
  - CHU St Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No